CLINICAL TRIAL: NCT02202668
Title: Transcutaneous Raman Spectroscope Analyses of Diabetic Foot Ulcers
Brief Title: Transcutaneous Raman Spectroscope (TRS) Analyses of Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: TRS probe performance does not meet primary outcome data requirements
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Blake Roessler, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00083401
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Foot Ulcer
Keywords: Foot ulcer, diabetic; Spectrum analysis, Raman
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRS (Experimental)
  Interventions: Device: TRS

INTERVENTIONS:
Device: TRS — TRS measurements of subcutaneous deep wound soft tissue and underlying bone will be collected at the same standard locations that are used to measure wound dimensions. The probe will never be in contact with the wound, but we will sterilize the probe head in advance in order to ease potential concerns regarding equipment sterility. A single point TRS measurement can be obtained in less than 60 seconds. At a minimum we will collect measurements at the geometric center of the wound as well as at the "6 and 12" and "3 and 9" ulcer coordinates. These coordinates are commonly used to estimate ulcer dimensions. It is anticipated that the PhAT probe will be used with a beam diameter of 7.5 mm. It is possible that the incident laser beam diameter will need to be adjusted (7.5 mm to 6.0 mm) to accommodate smaller wounds. If incident laser beam diameter adjustment is necessary we will also adjust the laser intensity to maintain the maximum permissible exposure of 0.3 W/cm2 per ANSI guidelines.

SUMMARY:
The primary translational research objective of the study is to demonstrate feasibility of using the Transcutaneous Raman Spectroscopy technology in a point-of-care environment. This study represents an initial evaluation of the device in a small cohort of human patients with diabetic foot ulcers. We will be evaluating safety, device design and certain human engineering factors associated with point of care use of the TRS. We anticipate the data we collect in this study will form the basis of later medical device studies.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Diagnosis of diabetes mellitus
* Full thickness or superficial foot and ankle ulcers based on clinical assessment (e.g., University of Texas (UT) grades 1-3, stages A-D). For reference, see Appendix 1 for the UT classification table

Exclusion Criteria:

* Age less than 18 or greater than 80 years old
* Subject has a psychological or sociological condition or an addictive disorder that would preclude informed consent
* Completely epithelialized ulcer based on clinical assessment with no ischemia or infection (UT classification 0A)
* Current or previous use of anti-resorptive bisphosphonate drugs (e.g., risedronate (Actonel) and alendronate (Fosamax))

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Transcutaneous Raman spectra of subcutaneous deep wound soft tissue and underlying bone | Baseline, then monthly for 3 months
  We will equip our portable Raman instrument with a non contact probe (PhAT probe, Kaiser Optical Systems). The probe will be placed ~ 10 inches from the wound and it will not be in contact with the wound. Depending on the size of the wound, the laser spot size on the wound bed will be 6-7.5 mm. The Raman spectra are derived from the laser light reflected back into the probe and captured by a charge coupled device (CCD) in the spectroscope. Computer software algorithms are used to deconvolute the CCD information into an interpretable Raman spectrum.

SECONDARY OUTCOMES:
Wound temperature post-Transcutaneous Raman Spectroscope | Baseline then monthly for 3 months
  Local temperature measurements of the wound will be collected before and immediately after the Raman measurements using a commercially available non-contact infrared thermometer which is also used to measure temperature in pediatric patients

CONTACTS AND LOCATIONS:
Overall Officials: Blake Roessler, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States